CLINICAL TRIAL: NCT05782335
Title: Analysis of T and B Cell Repertoire Changes and CTLA4 Genetics and Gene Expression to Understand the Mechanisms of Treatment Response to Orencia ® (Abatacept) in Rheumatoid Arthritis
Brief Title: Analysis of T and B Cell Repertoire Changes in Response to Orencia® (Abatacept) in Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0142
Record Dates: First submitted 2023-02-16; First posted 2023-03-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: abatacept; b cell repertoire; t cell repertoire
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample prior to infusion at all visits,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: Abatacept Initiator: RA patients of any disease duration, 18 years or older who are starting ABA (either IV or subcutaneous at standard doses) for the first time. Concomitant non-biologic medications (for e.g., standard conventional synthetic (cs)DMARDs, one of which must be MTX as typically used in routine care, or if MTX was not tolerated leflunomide will be acceptable) will be allowed as long as the dose has been stable for at least 3 months.
- Arm 2: csDMARD/TNFi Treated: RA patients, 18 years or older and on stable doses of conventional DMARDs (MTX with or without hydroxychloroquine, sulfasalazine, with or without leflunomide therapy, where leflunomide therapy can be an alternate to MTX). Patient's disease activity can be controlled or near controlled (CDAI <=12) or active if a recent DMARD or TNFi has been added, though they will have been on MTX at doses of at least 15mg weekly or leflunomide 10 mg or more for 4 weeks or more. A combination of csDMARDs at stable doses for 4 or more weeks with >= MTX 10 mg weekly or ± MTX 10 mg weekly for at least 4 weeks with any dose of a conventional TNF inhibitor (stable dose + TNFi) is permitted.
- Arm 3. Healthy Controls: Healthy individuals over 18 y.o. without RA, SLE, juvenile arthritis, psoriasis or psoriatic arthritis or other inflammatory auto-immune rheumatic disease, who are receiving care at the HSS or volunteers from the community. Participants will be recruited to serve in the control population for this study. Given that the range of age for most RA patients is between 40-70, we will aim to recruit control volunteers in this age range, ensuring that at least 60% - 70% are female, ensuring an age range and sex that is proportionately similar to the RA population at HSS.

SUMMARY:
The condition that will be studied is Rheumatoid Arthritis (RA), and in particular, RA patients with moderate to highly active disease who were prescribed Abatacept (Orencia®) (ABA) by their physician during their setting of care at Hospital for Special Surgery (HSS). This investigator-initiated, prospective, comparative, 3-arm observational study will examine changes in lymphocytes in RA patients starting abatacept compared to RA patients starting TNF inhibitors and to healthy controls. This will help investigators to learn more about the processes that cause joints to swell and hurt. This may also offer clues that might predict which patients will have a good or poor response to these treatments.

DETAILED DESCRIPTION:
This is a mechanistic study examining changes in repertoires of both T cell receptors (TCR) and B cell receptors (BCR) in patients with RA initiating ABA treatment and who are followed for 6 months relative to changes in repertoires of both TCRs and BCRs in two similarly followed comparator groups: . Patterns of T and B cell repertoires in the group of patients with RA initiating treatment with ABA will be compared to (i) RA patients on stable therapy with methotrexate (MTX) or leflunomide (LEF) with or without TNF inhibitors and (ii) "controls" matched for age (+/- 7 years) and sex (approximately 75% female +/- 5%). Our primary hypothesis is that ABA treatment will affect the immune repertoires both in TCR and BCR and the distribution of immune cell subsets (particularly B cell subsets) over time to a greater extent than non-ABA treated RA patients and "controls".

The goal is to determine how abatacept changes the repertoires of both TCRs and BRCs compared to control groups. The investigators anticipate that the repertoires will change differently in ABA treated patients over time relative to similar RA patients treated with conventional synthetic DMARDS (MTX and / or Leflunomide), with or without the use of a TNF inhibitor (TNFi). Changes in repertoires will also be compared to "controls" with no inflammatory disease.with proportionately similar proportions of anti-CCP3 positivity, (but not anti-IL-6 therapy, Jak Kinase Inhibitors (JAKi's) or Rituximab)

A total of 72 people will participate in this study at HSS in three separate arms:

* Arm 1: Patients beginning abatacept as a treatment for their RA
* Arm 2: Patients beginning a TNF inhibitor as a treatment for their RA
* Arm 3: Healthy volunteers (free from autoimmune or connective tissue disease)

Once enrolled, these participants will be assessed at their baseline visit and seen 3 months and 6 months after baseline. These visits will involve a blood draw and questionnaires related to functioning and feeling with RA (where applicable) and may take up to an hour. Participants will be compensated per visit.

ELIGIBILITY:
Inclusion Criteria: M or F >=18 y.o. with diagnosed RA. Disease related inclusion criteria:

1. Patients being treated with MTX with or without csDMARDS at stable doses for at least 4 weeks, who are either: (a) about to start ABA, OR, (b) who are likely to remain on stable DMARDs and who might also be using a TNFi but in whom all therapies will have been stable for 4 or more weeks.

2.) meet diagnostic criteria for RA, based on 2010 ACR Criteria or 1987 RA criteria, OR, are one point short of meeting the criteria but are being treated for RA, OR, have previously identified RA typical erosions.

3) have never received ABA or rituximab, and, if previously used a JAKi, will have stopped this for over a month, OR, if previously used an IL-6 inhibitor, will have stopped for at least 3 months.

4) RA subject must not be taking prednisone at doses over 10 mg daily, and will not have received injectable Depomedrol or equivalent within 4 weeks of baseline or prior to the 3 or 6 month study assessment. Healthy control patients cannot be taking prednisone. Any subject can use oral or nasal inhalers that include glucocorticoids 5) have evidence of recent or currently active disease depending on treatment arm. Subjects starting ABA (Arm 1) are expected to have at least moderate disease activity, OR if CDAI is between 2.81 and 10, there should be two or more swollen and tender joints. For subjects being included in Arm 2, the stable treatment arm, CDAI <13 and one swollen joint observed by a rheumatologist in the prior 6 months. Subjects recruited to the healthy control arm (Arm 3) will be free of any autoimmune disease or systemic form of an inflammatory arthritis.

6) WOCBP must be using acceptable forms of contraception to avoid pregnancy throughout the study, i.e. oral contraceptives, other hormonal contraceptives.

Specific Exclusion Criteria:

1. Have severe complications of RA that might require imminent escalation of therapy, e.g. pericarditis, active vasculitis of a major organ system.
2. Have an autoimmune disease or systemic inflammatory rheumatic disease (e.g., lupus erythematosus) that could confound T and B cell subset results
3. Have a concurrent serious medical disease (e.g., terminal malignancy)
4. Have a BMI indicating poor health (<18 or > 40)
5. Have received the following Prohibited Treatments and/or Therapies

   1. treatment with rituximab
   2. exposed to ABA or CTLA-4Ig
   3. exposed to any investigational drug within 28 days.
   4. received any live vaccines within 2 weeks prior to study start. Subjects cannot receive a live vaccine at any time during the study.
6. WOCBP with a positive pregnancy test on enrollment or prior to study start, OR who are unwilling or unable to use an acceptable method to avoid pregnancy despite continuing MTX.
7. part of a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is patients with RA who are starting ABA. Data from the study population will be compared with RA controls being treated with standard of care therapy, i.e., MTX with or without either other conventional synthetic (cs)DMARDs and/or a TNF inhibitor (etanercept, adalimumab, golimumab, infliximab, certolizumab pegol). RA patients who enter the study must meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in clonotype diversity of T cell and B cell repertoires | April 2024-March 2025
  Investigators will compare the change in clonotype diversity of T cell and B cell repertoires in patients over 6 months by analyzing clonotype diversity of T cell and B cell repertoires at BL (pre-treatment), 3 months, and 6 months post treatment for each individual in each of the three groups (RA starting ABA; RA on stable MTX +/- TNFi.

SECONDARY OUTCOMES:
CTLA4 gene expression in peripheral blood at 3 times points | April 2024-March 2025
  Investigators will assess changes in CTLA4 gene expression in peripheral blood at BL, and at 3 and 6 months post-treatment.
Changes in the proportions of T and B cell subtypes | April 2024-March 2025
  Changes in the proportions of T and B cell subtypes well as NK cells associated with ABA treatment. Flow cytometry analysis will be used to quantify the frequency of T and B cell subtypes and NK cells at each timepoint in each subject in each Arm.
Expression levels in peripheral blood of genes key to the immune response. | April 2024-March 2025
  Changes in expression levels in peripheral blood of 150 genes key to the immune response.

OTHER OUTCOMES:
T cell and B cell repertoire changes and CDAI | April 2024-March 2025
  Association between T cell and B cell repertoire changes and clinically meaningful improvements in CDAI.
T cell and B cell repertoire changes and SDAI. | April 2024-March 2025
  Association between T cell and B cell repertoire changes and clinically meaningful improvements in SDAI.
T cell and B cell repertoire changes and DAS23-ESR. | April 2024-March 2025
  Association between T cell and B cell repertoire changes and clinically meaningful improvements in DAS23-ESR.
T cell and B cell repertoire changes and DAS-28-CRP. | April 2024-March 2025
  Association between T cell and B cell repertoire changes and clinically meaningful improvements in DAS28-CRP.
RA-FQ in ABA treated vs. non-ABA treated patients | Aprill 2024-March2025
  Patient reported outcome (PRO) measure (RA-FQ) in ABA treated patients over 6 months compared to non-ABA treated RA patients.
MD-HAQ in ABA treated vs. non-ABA treated patients | Aprill 2024-March2025
  Patient reported outcome (PRO) measure (MDHAQ) in ABA treated patients over 6 months compared to non-ABA treated RA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bridges, MD PhD, Principal Investigator — Hospital for Special Surgery, New York; Vivian P Bykerk, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No